Date: September 1, 2021

Title: Comparison Effects Of Blue Prescription Program, Home Exercise Program And Supervised Exercise Approaches On Type 2 Diabetic Women.

Identifiers: NCT05479435

Statistical Analysis Plan

SPSS 22.0 for MacBook was utilized to analyze the data. The Shapiro-Wilk test was employed to assess whether the data exhibited a normal distribution. Mean, standard deviation, median, and frequency were provided for quantitative data and compared using ANOVA test. Chisquare test was applied for qualitative data analysis. ANCOVA test was utilized for intergroup comparisons of normally distributed data, and Tukey test was used for post hoc analyses. For intra-group comparisons, data were analyzed with paired t-test. Intergroup comparisons of nonnormally distributed data were conducted using the Kruskal-Wallis test, and intragroup comparisons were performed with the Wilcoxon signed-rank test. Mann-Whitney U test was employed for pairwise comparisons. The significance level was set at  $p \le 0.05$